CLINICAL TRIAL: NCT03133962
Title: Evaluation of the Contribution of the Ultrasound Tracking and the Positioning of the Distal End During the Implantation of Implantable Chamber or Long-lasting Venous Catheter
Acronym: EchoPAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of the investigator
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2014_843_0013
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Echocardiography; Implantable Chamber

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients applying for CAP or long-term central catheter (Other)
  Interventions: Other: Adult patients who are candidates for a CAP or long-term central catheter placement

INTERVENTIONS:
Other: Adult patients who are candidates for a CAP or long-term central catheter placement — Evaluate the feasibility of finding the correct positioning of the distal end of the PAC or of the long-term catheter by cardiac ultrasound in comparison with the brightness scopy, reference method.

SUMMARY:
Given the increase in the number of PAC implants or long-term catheters, and the ease of access to cardiac ultrasound in the operating theaters, the investigator thought to use ultrasound to PAC or long-term catheters.

The investigator considers cardiac echocardiography through its costal pathway to locate the correct positioning of the distal end of the catheter in a manner equivalent to the scopic locating with all the side effects of the irradiation and with Equivalent efficiency

ELIGIBILITY:
Inclusion Criteria:

* All adult patients are candidates for a long-term CAP or central catheter placement.
* Benefiting from sedation or general anesthesia.

Exclusion Criteria:

* Patient aged <18 years.
* Pregnant woman.
* Lack of anesthesiologist with knowledge of ultrasound.
* Site of femoral puncture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
Good positioning of the distal end of the catheter by ETT, without repositioning following the scopy | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France